CLINICAL TRIAL: NCT07307456
Title: A Prospective, Open-label, Single-center Clinical Study Evaluating the Efficacy and Safety of Trastuzumab Combined With BCG Perfusion as an Adjuvant Treatment After TURBT in High-risk/Very High-risk Non-muscle-invasive Bladder Cancer
Brief Title: Tremelimumab Combined With BCG Perfusion for the Treatment of HR-NMIBC After TURBT Surgery Exploration
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Shuxiong Zeng, associate chief physician, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTSB20250508008
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer
Keywords: HR-NMIBC; Immunotherapy; BCG; Bladder preservation treatment
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with toripalimab combined with BCG instillation after TURBT in patients with HR - NMIBC (Other)
  Interventions: Drug: Treatment with toripalimab combined with BCG perfusion following transurethral resection of bladder tumor (TURBT)

INTERVENTIONS:
Drug: Treatment with toripalimab combined with BCG perfusion following transurethral resection of bladder tumor (TURBT) — This study employs a fixed-dose combination regimen. All enrolled patients with high-risk/very high-risk NMIBC, following TURBT, first receive a single 2000mg gemcitabine intravesical instillation. Subsequently, they undergo synchronized combination therapy consisting of fixed-dose 240mg toripalimab via intravenous infusion (every 3 weeks for 8 cycles) paired with standard BCG intravesical instillation (6-week induction phase + maintenance phases at months 3 and 6). Treatment continues until completion of the planned cycles, disease progression, or unacceptable toxicity. The protocol includes detailed dose-modification guidelines for immune-related adverse events based on CTCAE v5.0.

SUMMARY:
This is a single-center, prospective, open-label, non-randomized clinical study initiated and conducted by the Department of Urology, Shanghai Changhai Hospital. The Principal Investigators are Professor Zhang Zhensheng and Professor Chen Guanghua. The projected study period is from December 2025 to December 2028. This study aims to evaluate the efficacy and safety of toripalimab (a PD-1 inhibitor) combined with Bacillus Calmette-Guérin (BCG) intravesical instillation as adjuvant therapy following transurethral resection of bladder tumor (TURBT) in patients with high-risk/very high-risk non-muscle-invasive bladder cancer (NMIBC).

Bladder cancer is a common malignancy of the urinary system, with NMIBC accounting for approximately 75% of initial diagnoses. For high-risk patients who are unresponsive to or experience recurrence after BCG therapy, radical cystectomy remains the standard treatment. However, this procedure is associated with high rates of complications, mortality risk, and significantly negative impacts on quality of life. Therefore, exploring novel combination strategies that effectively reduce recurrence while preserving the bladder is of great clinical importance. This study is based on the successful application of immune checkpoint inhibitors in advanced urothelial carcinoma and recent Phase III trials (e.g., the CREST study) demonstrating the efficacy and safety of combining PD-1/PD-L1 inhibitors with BCG in treatment-naïve high-risk NMIBC. It seeks to investigate the potential of the domestic PD-1 inhibitor toripalimab in combination with standard BCG instillation.

The study plans to enroll 31 patients with histologically confirmed high-risk/very high-risk NMIBC who have not previously received immune checkpoint inhibitors or BCG therapy. All enrolled patients will first receive a single instillation of gemcitabine (2000mg), followed by the combination therapy phase: toripalimab (240mg, intravenous infusion, every 3 weeks for 8 cycles) combined with BCG intravesical instillation (induction phase for 6 weeks, maintenance phases at months 3 and 6). The primary efficacy endpoint is the pathological complete response (CR) rate at approximately 6 months after treatment initiation. Secondary efficacy endpoints include duration of CR, 6-month and 2-year event-free survival (EFS) rates, 1-year and 2-year cancer-specific survival (CSS) rates, time to radical cystectomy, and overall survival (OS). Safety endpoints encompass the incidence and severity of adverse events (AEs) and serious adverse events (SAEs).

Statistical analyses will be based on the Full Analysis Set (FAS) and Per-Protocol Set (PPS). The sample size calculation for the primary endpoint (6-month CR rate) is based on historical data assumptions, employing a one-sided test. Safety analyses will include all patients who received at least one dose of study treatment. This study will strictly adhere to the principles of the Declaration of Helsinki, Chinese Good Clinical Practice (GCP) guidelines, and relevant regulations. The study protocol has been submitted for review and approval by the Institutional Review Board (IRB)/Ethics Committee. Written informed consent will be obtained from all patients prior to participation. This study aims to provide a new and potentially more effective bladder-preserving treatment option for patients with high-risk/very high-risk NMIBC and to evaluate the safety profile of this combination regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Patients with a pathological diagnosis of high-risk or very high-risk non-muscle-invasive bladder cancer (NMIBC) following transurethral resection or cystoscopic biopsy.

"High-risk patients" must meet any one of the following criteria:

1. All T1 high-grade (HG)/G3 without carcinoma in situ (CIS), excluding those in the very high-risk group.
2. All CIS patients, excluding those in the very high-risk group.
3. Ta low-grade (LG)/G2 or T1 G1 without CIS, accompanied by three risk factors.
4. Ta HG/G3 or T1 LG without CIS, accompanied by at least two risk factors.
5. T1 G2 without CIS, accompanied by at least one risk factor. "Very high-risk patients" must meet any one of the following criteria:

(1) Ta HG/G3 with CIS accompanied by three risk factors. (2) T1 G2 with CIS accompanied by at least two risk factors. (3) T1 HG/G3 with CIS accompanied by at least one risk factor. (4) T1 HG/G3 without CIS, accompanied by three risk factors. (Risk factors: age >70 years; tumor diameter >3 cm; multiple papillary carcinomas) 3. No prior treatment with therapies targeting PD-1, PD-L1, PD-L2, or CTLA-4, or other antibodies or drugs specifically targeting T-cell co-stimulation or checkpoint pathways (immune checkpoint blockers), or bacille Calmette-Guérin (BCG) therapy.

4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. 5. Adequate organ function, defined as meeting the following criteria (within 14 days prior to enrollment, without transfusion or granulocyte colony-stimulating factor treatment): "Hematology": i. Absolute neutrophil count (ANC) ≥1,000/mm³ ii. Platelet count ≥75,000/mm³ iii. Hemoglobin ≥8.0 g/dL "Hepatic function": i. Total bilirubin ≤1.5 × upper limit of normal (ULN) OR direct bilirubin ≤ ULN for subjects with total bilirubin >1.5 × ULN.

ii. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN.

"Renal function": Creatinine clearance (CrCl) >30 mL/min, calculated using the Cockcroft-Gault formula.

6. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to enrollment, be willing to use effective contraception during the study period and for at least 6 months after the last dose of study drug (including chemotherapy agents and toripalimab). Male subjects with female partners of childbearing potential must agree to use effective contraception during the study period and for at least 6 months after the last dose.

7. Subjects voluntarily agree to participate in the study by providing written informed consent, demonstrate good compliance, and are willing to cooperate with follow-up.

Exclusion Criteria:

Patients meeting any of the following criteria were excluded from this study:

1. History or presence of muscle-invasive or disseminated/metastatic bladder cancer. Patients with locally advanced or metastatic bladder cancer or concurrent upper tract urothelial carcinoma were excluded.
2. Prior surgical intervention for bladder cancer other than transurethral resection of bladder tumor (TURBT) and/or bladder biopsy.
3. Administration of any other approved systemic anticancer therapy or systemic immunomodulatory agents (including, but not limited to, interferon, interleukin-2, and tumor necrosis factor) within 28 days prior to enrollment.
4. Severe chronic or active infection requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days prior to enrollment.
5. Major surgery or significant trauma within 28 days prior to enrollment.
6. Vaccination with a live vaccine within 28 days prior to enrollment.
7. Use of any Chinese herbal medicine or proprietary Chinese medicine for cancer control within 14 days prior to enrollment.
8. Treatment with systemic corticosteroids within 4 weeks prior to the study intervention.
9. Active autoimmune diseases requiring systemic treatment or other conditions necessitating long-term use of high-dose corticosteroids and other immunosuppressive agents.
10. History of potassium, sodium, or calcium abnormalities, hypoalbuminemia, interstitial lung disease, non-infectious pneumonitis, or other uncontrolled systemic diseases (including diabetes, hypertension, cardiovascular diseases, etc.) that, in the investigator's judgment, could affect the treatment.
11. Active viral hepatitis B or C. Patients with acute or chronic active hepatitis B or C infection were excluded if they met any of the following criteria: hepatitis B virus (HBV) DNA >2000 IU/mL or 10⁴ copies/mL; hepatitis C virus (HCV) RNA >10³ copies/mL; or co-positivity for hepatitis B surface antigen (HBsAg) and anti-HCV antibody.
12. Known history of human immunodeficiency virus (HIV) infection or known diagnosis of acquired immunodeficiency syndrome (AIDS) (no screening tests were required).
13. History of any organ transplantation, including allogeneic stem cell transplantation, except for transplants not requiring immunosuppression (e.g., corneal transplant, hair transplant).
14. Known history of allergic reactions to any of the study drugs.
15. Concurrent participation in another clinical trial.
16. History and/or concurrent presence of other malignancies, except for: malignancies treated with curative intent with no recurrence for over 3 years, or early-stage cancers considered cured, including completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.
17. Active central nervous system metastases or carcinomatous meningitis.
18. Any condition that, in the investigator's opinion, rendered the patient unsuitable for study participation (e.g., treatment not in the patient's best interest, poor patient compliance, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-12-08 (Estimated); Study Completion 2028-12-08 (Estimated)

PRIMARY OUTCOMES:
Six - month pathological complete remission (CR) rate | From the first administration of the investigational drug to six months after the treatment.
  (assessed via cystoscopy and urine cytology approximately six months after the first administration of the study drug)

CONTACTS AND LOCATIONS:
Locations (1):
- ChangHai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No